CLINICAL TRIAL: NCT03573128
Title: Development and Pilot Testing of the Students With Autism Accessing General Education (SAAGE) Model
Acronym: SAAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: May Institute (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Suzannah Iadarola, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A150032
Record Dates: First submitted 2018-06-06; First posted 2018-06-29 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Students with Autism Accessing General Education (SAAGE). Teaching staff work with a study team coach to identify areas of concern for individual students, create goals and implement a modular behavioral intervention using an active teaching/feedback loop model.
  Interventions: Behavioral: Students with Autism Accessing General Education
- Enhanced Services As Usual (Active Comparator): Teaching staff access in-service training sessions hosted by study team and are provided with print materials from which the modules for the active intervention were created.
  Interventions: Other: Enhanced Services As Usual

INTERVENTIONS:
Behavioral: Students with Autism Accessing General Education — With study team coach support, teacher implemented modules addressing student behavioral/academic goals.
  Arms: Intervention
Other: Enhanced Services As Usual — Teaching staff access in-service presentations and print materials with no active study team coaching.
  Arms: Enhanced Services As Usual

SUMMARY:
Study personnel will use evidence based behavioral skills training procedures to coach educators to implement modules designed to increase the quality of educational services and access to inclusive settings in elementary school for students with Autism Spectrum Disorder.

DETAILED DESCRIPTION:
This project brings together the expertise of investigators at three centers to develop and conduct a pilot test of a new comprehensive intervention to increase the quality of educational services and access to inclusive settings for students with autism spectrum disorder (ASD) in elementary school (kindergarten through 5th grade). The intervention model, Students with Autism Accessing General Education (SAAGE), integrates evidence-based strategies to teach skills to students with ASD in schools, best practices derived from this literature by the project investigators, a recent guidebook written by the principal investigator, and research on collaboration with community providers such as school teams to implement interventions efficaciously and sustainably. SAAGE begins with strategies to help a school form a cohesive team to oversee implementation of the model in the school. For each student, SAAGE uses a modular approach for identifying goals for a student, selecting appropriate teaching strategies, and systematically monitoring progress and trouble-shooting. The modules center on core and associated features of ASD. Study personnel will use well established behavioral skills training procedures to coach educators to implement the modules.

ELIGIBILITY:
Inclusion Criteria:

Children subjects:

* Are enrolled in school grades kindergarten through 5th
* Have an IEP educational classification of Autism, confirmed by the Autism Diagnostic Observation Schedule, Second Edition, and DSM-5 checklist
* No planned changes in school placement or core team members during the school year of participation

Adult subjects (teachers, para educators):

* Instructional personnel who currently support a participating child with ASD at school (e.g., teacher, instructional assistant, speech pathologist, occupational therapist)
* Letter from instructional personnel's district or school indicating agreement to take part in the research project

Exclusion Criteria:

Children subjects • Diagnosis of (1) genetic disorders such as Fragile X, Down syndrome, or tuberous sclerosis; 2) profound vision or hearing loss; or (3) motor disabilities such as cerebral palsy (these multiple disabilities would prevent standard implementation of the intervention protocol).

Adult subjects

• Instructional personnel whose written consent was not obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Mean change in student function as measured by the Developmental Disability-Clinical Global Assessment Scale | baseline to end of school year (approx. 9 months)
  The Developmental Disability-Clinical Global Assessment Scale ranges from 1-100 with 100 indicating superior functioning. It assesses student function in a classroom setting.

SECONDARY OUTCOMES:
Mean change in social communication and interaction as rated by child's teacher using the 30 item Social Skills Subscale of the Social Skills Improvement System | baseline to end of school year (approx. 9 months)
  The Social Skills Improvement System, Social Skills Subscale is a 30 item measure of social communication and interaction using a 4 point Likert scale to rate the frequency of behaviors and a 3 point Likert scale to the the importance of each item.
Mean change in restricted and repetitive behavior as measured by the Children's Yale-Brown Obsessive-Compulsive Scales - PDD | baseline to end of school year (approx. 9 months)
  The Children's Yale-Brown Obsessive-Compulsive Scales - PDD is a modified version of the Children's Yale-Brown Obsessive-Compulsive Scales which is adapted for use with children with ASD. It is a semi structured clinician rated scale designed to rate the current severity of repetitive behavior. Each item is scored on a 5 point scale from 0 to 4 with 4 being most symptomatic.
Change in teacher-nominated target behaviors | baseline to end of school year (approx. 9 months)
  Teacher Nominated Target Behaviors
Change in on-task behavior during instruction | baseline to end of school year (approx. 9 months)
  Academic Engaged Time
School-related adaptive functioning | baseline to end of school year (approx. 9 months)
  Adaptive Behavior Assessment System, Self-Direction Scale
Social skills and behavior regulation | baseline to end of school year (approx. 9 months)
  Social Skills Improvement System
Class placement | baseline to end of school year (approx. 9 months)
  IEP review

CONTACTS AND LOCATIONS:
Overall Officials: Tristram H Smith, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No